CLINICAL TRIAL: NCT03939273
Title: Randomized Placebo-controlled Study on the Effects of Antibiotic-induced Gut MicrobiomE Disruption on the Innate Immune Response Following Cardiac Surgery
Brief Title: The Effects of Gut Micribiota Disruption on the Immune Response After Open Heart Surgery
Acronym: REMEDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The REMEDI trial; 2019-000964-54 (EudraCT Number)
Record Dates: First submitted 2019-04-04; First posted 2019-05-06 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Systemic Inflammatory Response Syndrome; Postoperative Shock; Coronary Artery Disease; Extracorporeal Circulation; Complications
Keywords: Systemic Inflammation; Microbiome; CABG; Coronary Artery Bypass Graft; Innate Immunity; Gut microbiota
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Coronary Artery Disease | interventions — Vancomycin; Metronidazole; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): A preoperative seven day course of oral ciprofloxacin 500 mg twice a day, oral vancomycin 500 mg thrice per day, oral metronidazole 500 mg thrice per day and a six day course of oral fluconazole 200 mg once per day.
  Interventions: Drug: Vancomycin Oral; Drug: Metronidazole Oral; Drug: Ciprofloxacin Pill; Drug: Fluconazole Oral Product
- Control group (Placebo Comparator): A preoperative seven day course of placebo, consisting of pills and capsules identical in appearance and number to the active group
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Vancomycin Oral — 500 mg thrice per day for seven days
  Arms: Active group
Drug: Metronidazole Oral — 500 mg thrice per day for seven days
  Arms: Active group
Drug: Ciprofloxacin Pill — 500 mg twice per day for seven days
  Arms: Active group
Drug: Fluconazole Oral Product — 200 mg once per day for six days
  Arms: Active group
Drug: Placebos — seven day course of placebo tablets and capsules identical in appearance and number to active treatment
  Arms: Control group

SUMMARY:
In this randomized, double-blind, placebo-controlled study, the investigators will assess whether preoperative disruption of the gut microbiota by a course of broad spectrum antibiotics will attenuate the postoperative systemic inflammatory response after on-pump cardiac surgery

DETAILED DESCRIPTION:
During cardiac surgery, the use of cardiopulmonary bypass and extracorporeal circulation, operative trauma, and ischemia-reperfusion injury can induce a profound systemic innate immune response. This response contributes to postoperative morbidity and mortality, as increased proinflammatory cytokine levels are associated with several postoperative complications. Commensal microbiota in the gut can modulate systemic immune responses. The investigators hypothesize that reduction of systemic immune activation by disruption of the microbiome may be beneficial in patients undergoing cardiac surgery.

The objective of this trial is to assess the anti-inflammatory effects of disruption of the intestinal microbiota with broad-spectrum antibiotics in patients with systemic inflammation following cardiac surgery and to assess the effects on clinical outcomes in these patients.

To this end, subjects will be randomized into one of two treatment arms and will receive either active treatment or a placebo during the seven days prior to surgery. Active treatment consists of a seven day course of oral ciprofloxacin 500 mg twice a day, oral vancomycin 500 mg thrice per day, oral metronidazole 500 mg thrice per day and a six day course of oral fluconazole 200 mg once per day. Placebo treatment is randomly allocated in a double blind fashion in a 1:1 proportion to the active treatment. Stool samples will be obtained prior to and directly after study treatment to assess the effects on the richness and diversity of the gut microbiota. During and after surgery, plasma levels of circulating cytokines will be measured to assess the effects of microbiota disruption on the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Scheduled for elective on-pump cardiac surgery.
* Written informed consent to participate in this trial prior to any study-mandated procedure

Exclusion Criteria:

* Use of any antibiotic or antifungal therapies within 30 days prior to surgery
* History of inflammatory bowel disease
* History of bowel resection and / or short bowel syndrome
* Pre-operative creatinine clearance < 50 ml/min
* Severe hepatic impairment
* Immune compromised

  * Solid organ transplantation
  * Known HIV
  * Pregnancy
  * Use of immunosuppressive drugs
* Emergency surgery
* Haematological disorders

  * Disorders from myeloid and / or lymphoid origin
  * Leucopenia
* Known hypersensitivity to any of the investigational and/or non-investigational products or their excipients.
* Treatment with investigational drugs or participation in any other intervention clinical trial within 30 days prior to study drug administration
* Inability to personally provide written informed consent
* Suspected of not being able to comply with the trial protocol
* Use of vitamin K antagonists
* Use of tricyclic antidepressants
* Use of other drugs which have potential dangerous interactions with study treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Between group differences in Area Under the Curve (AUC) of the time-concentration curve of interleukin (IL)-6 plasma concentrations. | During surgery and up to 24 hours after surgery
  Blood samples will be obtained at predefined time points during and after surgery to assess plasma levels (in pg/mL) of circulating inflammatory mediators. To assess between group differences, the AUC of the time-concentration curve (expressed in arbitrary units) of each inflammatory mediator will be calculated.

SECONDARY OUTCOMES:
Between group differences in AUC of the time-concentration curve of other inflammatory mediators. | During surgery and up to 24 hours after surgery
  Tumor Necrosis Factor (TNF)-α, IL-8, IL-10, IL-1β, IL-1RA, Monocyte Chemoattractant Protein (MCP)-1, Macrophage Inflammatory Protein (MIP)-1α MIP-1β, Vascular Cell Adhesion Molecule (VCAM), Intercellular Adhesion Molecule (ICAM)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided